CLINICAL TRIAL: NCT00718094
Title: A Phase IIa Pilot Study to Determine the Safety of an Oral Dose of Green Tea Extract (Polyphenon E®) and Provide Preliminary Evidence to Support Its Efficacy in Ulcerative Colitis
Brief Title: Pilot Study of Green Tea Extract (Polyphenon E®)in Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gerald W. Dryden, Jr., Principal investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 390.05; 5K23DK073750 (NIH)
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Mild to Moderately Active Ulcerative Colitis
Keywords: Ulcerative colitis; EGCG; Green tea polyphenols; Inflammatory bowel disease; Colitis; IBD; Green tea
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Colitis | interventions — polyphenon E

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polyphenon E treatment (Experimental): Polyphenon E® therapy was given for 56 days.
  Interventions: Drug: Polyphenon E®
- Placebo (Placebo Comparator): Oral Placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Polyphenon E® — Oral capsules
  Arms: Polyphenon E treatment
Drug: Placebo Oral Tablet — Oral tablet: placebo
  Arms: Placebo

SUMMARY:
Green tea consists of several components, with most research focusing on the polyphenol fraction. The polyphenol fraction(-)-epigallocatechin-3-gallate (EGCG)has been studied extensively as an anti-inflammatory agent as well as a preventative agent for cancer. It has been shown to effectively reduce the inflammation associated with animal models of inflammatory bowel disease. This clinical trial will determine the ability of EGCG, in the form of Polyphenon E®, to treat patients with mild to moderately severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female with mildly to moderately active ulcerative colitis

Exclusion Criteria:

* Off prohibited medications for proscribed period of time
* Evidence of infectious colitis
* Labs outside of range
* Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald W Dryden, MD, MSPH, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Clinical Research Center, Louisville, Kentucky, United States

REFERENCES:
- [Result] Dryden GW, Lam A, Beatty K, Qazzaz HH, McClain CJ. A pilot study to evaluate the safety and efficacy of an oral dose of (-)-epigallocatechin-3-gallate-rich polyphenon E in patients with mild to moderate ulcerative colitis. Inflamm Bowel Dis. 2013 Aug;19(9):1904-12. doi: 10.1097/MIB.0b013e31828f5198. PMID 23846486

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyphenon Treatment: Polyphenon E®: Oral capsules for 56 days
Period: Overall Study
Arm/Group | Polyphenon Treatment | Placebo
Started | 15 | 5
Completed | 15 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polyphenon E Treatment | Placebo | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (15) | 30.7 (14.4) | 40 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 15 | 5 | 20
Ulcerative colitis (UC) disease activity index [Mean (Standard Deviation); unit: units on a scale] — This is a standard method of measuring disease activity. The index assesses four variables, which include stool frequency, severity of bleeding, colonic mucosal appearance, and the physician's overall assessment of disease activity.
  Each variable is scored from 0-3 so that the total index score ranges from 0-12; 0-2: remission; 3-6: mild; 7-10: moderate; >10: severe UC.
  units on a scale | 6.5 (1.7) | 7.3 (1.7) | 7.0 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Reduction in the Disease Activity Index of >3, or Clinical Remission.
Description: This Index is a measure of ulcerative colitis severity. The index assesses four variables, which include stool frequency, severity of bleeding, colonic mucosal appearance, and the physician's overall assessment of disease activity.
  Each variable is scored from 0-3 so that the total index score ranges from 0-12; 0-2: remission; 3-6: mild; 7-10: moderate; >10: severe UC.
Time Frame: day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Polyphenon E Treatment | Placebo
Number analyzed (Participants) | 15 | 5
Participants | 10 | 0
Statistical Analysis 1: Comparison: Polyphenon E Treatment vs Placebo; Test type: Superiority; p = 0.03, Fisher Exact

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Polyphenon E Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyphenon E Treatment (N=15) | Placebo (N=5)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes